CLINICAL TRIAL: NCT01209793
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study of the Safety and Tolerability of Intravenously Administered REGN846 (SAR302352) in Healthy Volunteers
Brief Title: Safety and Tolerability Study of REGN846 (SAR302352) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R846-HV-1007
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose 1 (Experimental): (3:1, active: placebo)
  Interventions: Biological: REGN846
- Dose 2 (Experimental): (3:1, active: placebo)
  Interventions: Biological: REGN846
- Dose 3 (Experimental): (3:1, active: placebo)
  Interventions: Biological: REGN846
- Dose 4 (Experimental): (3:1, active: placebo)
  Interventions: Biological: REGN846
- Dose 5 (Experimental): (3:1, active: placebo)
  Interventions: Biological: REGN846

INTERVENTIONS:
Biological: REGN846 — 5 IV cohorts (Dose 1, 2, 3, 4, 5)

SUMMARY:
This study is being conducted to assess the safety and tolerability of a single ascending intravenous (IV) dose of REGN846 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 18 and 65; women must be postmenopausal or surgically sterile
* Body Mass Index (BMI) between 18.0 and 30.0 kg/m2, inclusive
* Normal vital signs after resting in a sitting position for 5 minutes:
* Normal standard 12-lead ECG
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent
* Able to understand and complete study-related questionnaires

Exclusion Criteria:

* Current or prior history of smoking
* Any illness or condition that would adversely affect the subject's participation in this study
* Hospitalization within 60 days of the screening visit
* Any clinically significant abnormalities observed during the screening visit
* History of or positive human immunodeficiency virus (HIV) screen result at the screening visit
* History of positive blood test for hepatitis B/hepatitis C or positive hepatitis screen result at the screening visit
* History of positive drug screen result for drug or alcohol abuse within a year prior to the screening visit
* Known sensitivity to any of the components of the Investigational Product formulation
* Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit
* Any condition that would place the subject at risk, interfere with participation in the study
* History of a parasitic infection or recent (within the previous 6 months) travel to a parasitic endemic area
* Live/attenuated vaccinations within 12 weeks of screening or during the study
* Any subjects with planned elective surgery
* Sexually active men who are unwilling to utilize adequate contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Baseline through end of study

SECONDARY OUTCOMES:
PK profile | Baseline through end of study
Immunogenicity | Visits 2, 8, 10 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Nucleus Network, Melbourne, Australia